| 1 | SUCCESSFUL TRANSITION FROM INSULIN PUMP TO MULTIPLE DAILY |
|----------|------------------------------------------------------------------|
| 2 3 | INJECTIONS USING INSULIN DEGLUDEC IN ADULTS WITH TYPE 1 DIABETES |
| 3 | (TRANSITION CLINICAL TRIAL) |
| 4 | |
| 5 | |
| 6 | |
| 7 | |
| 8 | INVESTIGATOR-SPONSORED STUDY PROPOSAL |
| 9 | |
| 10 | UNIVERSAL TRIAL NUMBER (UTN) |
| 11 | (U1111-1214-1853) |
| 12 | |
| 13 | CINICAL TRIAL NUMBER: NCT03987191 |
| 14 | |
| 15 | |
| 16 | |
| 17 | |
| 18<br>19 | |
| 20 | Barbara Davis Center for Diabetes |
| 21 | University of Colorado Denver |
| 22 | 1775 Aurora Ct, Room M20-1318 |
| 23 | Aurora, CO 80045 |
| 24 | Traidia, Co ooo is |
| 25 | |
| 26 | |
| 27 | <u>Correspondence</u> |
| 28 | |
| 29 | Viral Shah, MD |
| 30 | Assistant Professor of Medicine & Pediatrics |
| 31 | Barbara Davis Center for Diabetes, Adult Clinic |
| 32 | School of Medicine |
| 33 | University of Colorado Anschutz Medical Campus |
| 34 | 1775 Aurora Ct, Room M20-1318 |
| 35 | Aurora, CO 80045 |
| 36 | Phone:303-724-8186 |
| 37 | Fax: 303-724-6784 |
| 38 | viral.shah@cuanschutz.edu |
| 39 | |
| 40 | |
| 41 | |
| 42 | |
| 43 | |

| <ul><li>44</li><li>45</li></ul> | | | Table of contents |
|---|---|---|---|
| 46<br>47 | 1. | BACI | KGROUND AND SIGNIFICANCE:4 |
| 48 | 2. | SPEC | CIFIC OBJECTIVES:6 |
| 49 | 3. | RESE | EARCH DESIGN AND METHODS:6 |
| 50 | | 3.1. | Study Hypothesis |
| 51 | | | Endpoints: |
| 52 | | 3.3. | Study design: |
| 53 | | | Rationale for study design |
| 54 | 4. | | ICAL RESEARCH SITES9 |
| 55 | 5. | STUI | DY POPULATION: |
| 56 | | 5.1. | Inclusion criteria |
| 57 | | 5.2. | Exclusion criteria |
| 58 | | 5.3. | Withdrawal criteria |
| 59 | | 5.4. | Subject replacement |
| 60 | | 5.5. | Rationale for study population |
| 61 | 6. | VISIT | T PROCEDURES: 13 |
| 62 | | 6.1. | Visit 1, screening and blinded CGM insertion |
| 63 | | 6.2. | Screening Failure |
| 64 | | 6.3. | Visit 2, Randomization visit |
| 65 | | 6.4. | Phone call 1 and phone call 2 |
| 66 | | 6.5. | Visit 3, end of treatment |
| 67 | | 6.6. | Phone call 3, follow-up phone call and end of the study |
| 68 | | 6.7. | Table 4: study visit outline |
| 69 | | 6.8. | Assessments for Safety: 23 |
| 70 | | 6.9. | Assessments for Efficacy: 23 |
| 71 | 7. | EVAl | LUABILITY OF SUBJECTS: |
| 72 | 8. | STAT | TISTICAL CONSIDERATIONS: 23 |
| 73 | | 8.1. | Sample size calculation |

| 74 | | 8.2. Statistical Methods | 25 |
|---|---|---|---|
| 75 | 9. | DATA HANDLING AND RECORD KEEPING: | 26 |
| 76 | 10. | ETHICS: | 27 |
| 77 | 11. | STUDY SCHEDULE: | 28 |
| 78 | 12. | STUDY DRUGS AND MATERIALS: | 28 |
| 79 | | 12.1. Study medications(s) / device(s) | 28 |
| 80 | | 12.2. Packaging and labelling of study medication(s) | 29 |
| 81 | | 12.3. Storage and drug accountability of study medication(s) | 29 |
| 82 | | 12.4. Auxiliary supply | 30 |
| 83 | 13. | CONCOMITANT ILLNESS(ES) AND MEDICATION(S) | 30 |
| 84 | 14. | ADVERSE EVENTS: | 30 |
| 85 | | 14.1. Precautions/over-dosage | 36 |
| 86<br>87 | 15. | 14.2 Risks and Discomforts | |
| 88 | 16. | REFERENCES: | 40 |
| 89<br>90<br>91<br>92<br>93<br>94 | 17.<br>18. | Appendix 1Protocol Changes | |
| 95 | | | |
| 96 | | | |
| 97 | | | |
| 98 | | | |
| 99 | | | |
| 100 | | | |
| 101 | | | |
| 102 | | | |
| 103 | | | |
| 104 | | | |

106

107

108

109

110

111

112

113

114

115

116

117

118

119

120

121

122

123

124

125

126

| 1. | BACKGROUND | AND SIGNIFICANCE: |
|----|------------|-------------------|
|----|------------|-------------------|

Type 1 diabetes (T1D) is an autoimmune disease characterized by loss of insulin-producing pancreatic beta cells [1]. Patients with T1D require lifelong insulin therapy to maintain good glycemic control and reduce the risk for microvascular complications [2].

Despite many advances in insulin delivery methods, recent data from the Type 1 Diabetes Exchange Clinic Registry showed that only about 50% of people with T1D are using an insulin pump (continuous subcutaneous insulin infusion, CSII) as their insulin delivery method [3,4]. In addition, the overall frequency of pump discontinuation is 3%, being higher in adolescents (4%) and young adults (4%) than in young children (3%) or older adults (1%) [5]. Reasons behind pump therapy discontinuation, either after a short- or long- standing usage, can be different. The most commonly reported ones are issues with wearability, including problems with insertion, pump discomfort, skin reactions, adhesive problems, and interference with sports and activities. Other common ones included the feeling of anxiety, discontinuation recommended by health care practitioner, failure with glycemic control and pump working properly (i.e. infusion set failure) [5,6]. Moreover, many T1D patients on CSII treatment often go on a "pump vacation", periods of the year during which the patient decides to temporarily go back on multiple daily insulin injections (MDI). Reasons for taking a pump vacation can be very different, the most common ones being related to esthetic reasons (i.e. during summer period at the seaside) and during holidays [7].

Insulin degludec is a new ultra-long acting insulin. To date, it is the only insulin analogue to self-associate into multi-hexamers upon subcutaneous injection, resulting in a soluble depot from

which it is slowly and continuously absorbed into the circulation [8-9]. In the pharmaceutical formulation, i.e. in the presence of phenol and zinc, the insulin degludec hexamers adopt a conformation where only one of the ends is available to interact with the side chain of another hexamer and thus forms stable di-hexamers. Upon diffusion of phenol following injection, the insulin degludec di-hexamers open at both ends and lead to the formation of multi-hexamers. The gradual diffusion of zinc from the ends of the multi-hexamers causes terminal insulin degludec monomers to slowly and steadily dissociate, resulting in a slow and gradual delivery of insulin degludec from the subcutaneous injection site into the circulation [8-10]. This is the major difference with insulin glargine which, following subcutaneous injection, forms microprecipitates that must re-dissolve prior to absorption and which renders its absorption inherently variable [8-10].

The longer duration of action and the lower day-to-day insulin degludec variability makes it an appealing choice when patients want to start multiple daily injections. In addition, when compared to insulin glargine, insulin degludec is associated with lower incidence of nocturnal and overall hypoglycemia in insulin requiring patients with diabetes [11].

However, differently from insulin glargine, the time needed from first dose of insulin degludec to reach steady state, defined as serum concentration exceeding 90% of the final plateau, is about 2 to 3 days, being at 60% of steady state within at day 1 and 85% at day 2 [12-13]. This results in an increased risk of hyperglycemia, during the initial 48-72 hours of CSII to MDI transition using insulin degludec.

Current CSII to MDI transition strategy is to stop CSII and initiate long acting insulin (such as glargine or detemir 1:1) from day 1 of stopping insulin pump [14-17]. However, the standard of care strategy has not been successful at the Barbara Davis Center for Diabetes, a leading T1D center in the world (unpublished observation), due to significant hyperglycemia during the first 48-72 hours of this transition. Hyperglycemia for initial 2-3 days makes transition from CSII to MDI difficult and frustrating for the patients. Therefore, there is a need to have a standardized approach to transitioning patients from CSII to MDI using insulin degludec.

Considering the lack of evidence and knowledge gap, this study is proposed to examine an investigational approach in contrast to the clinical standard of 1:1 dose conversion in an attempt to lower the incidence and/or duration of hyperglycemia after transition from insulin pump.

## 2. SPECIFIC OBJECTIVES:

- 158 The primary objective of this study is to evaluate the efficacy and safety of an alternative CSII to
- MDI transition strategy using insulin degludec compared to the standard of care in adults with
- 160 T1D.

147

148

149

150

151

152

153

154

155

156

157

## 161 3. RESEARCH DESIGN AND METHODS:

- 162 3.1. Study Hypothesis
- We hypothesize that, as compared to the actual standard of care transition strategy (1:1 dose
- 164 conversion at the day of CSII to MDI transition), an alternative transition strategy will result in
- lower time spent in hyperglycemia without increasing the risk for hypoglycemia. The alternative
- strategy being (overlap transition strategy):
- Administration of insulin degludec at a 1:1 basal dose conversion dosage at day 0, with the concomitant use of the insulin pump for 48 hours from transition, where CSII basal rate

| 169 | | will be reduced by 50% during the first 24 hours from transition and by 75% during 24 to |
|---|---|---|
| 170 | | 48 hours from transition. CSII will be disconnected after 48 hours from transition. |
| 171 | 3.2. E | ndpoints: |
| 172 | Prima | ry and secondary endpoints will be analyzed from 1-week of blinded CGM use during |
| 173 | rando | mization phase. |
| 174 | Prima | ry endpoint: |
| 175 | 1. | Time spent in CGM glucose levels >180mg/dl |
| 176 | Secon | dary endpoints: |
| 177 | 1. | Time spent in CGM-measured "time-in-range" (glucose levels ≥70 mg/dl and ≤180 mg/dl) |
| 178 | 2. | Time spent in CGM-measured hypoglycemia < 70 mg/dl |
| 179 | 3. | Frequency of severe hypoglycemia as defined by the ADA (severe cognitive impairment |
| 180 | | requiring external assistance for recovery) and severe hyperglycemia (BG\ge 250 needing |
| 181 | | hospitalization) |
| 182 | 4. | Number of boluses (correction boluses) between groups during first 72 hours of |
| 183 | | randomization |
| 184 | 5. | Patient-Reported Outcomes (PRO) using validated questionnaires; insulin delivery |
| 185 | | satisfaction survey (IDSS) and Work Productivity and Activity Impairment Questionnaire: |
| 186 | | Specific Health Problem V2.0 (WPAI: SHP) [18,19] |
| 187 | 3.3. S | tudy design: |
| 188 | • | This is a 3-week, randomized control, open label, single center clinical trial with two study |
| 189 | | arms comparing the efficacy and safety of the 'standard of care transition' and an 'overlap |

transition' strategy

- The study consists of a screening phase, one week of run-in phase (blinded CGM monitoring), one week of the experimental protocol following randomization phase and one week of follow-up phase.
- Overall, the study will last 3 weeks that includes four clinical trial phases (**Figure 1**):
  - Screening phase (Week 0): After informed consent, inclusion and exclusion, blinded CGM
     will be inserted.
  - Run-in phase (Week 0 to end of week 1): Subjects will wear blinded CGM and continue to use CSII.
  - o <u>Randomization phase</u> (Week 1 to week 2): Subjects will be randomly allocated to one of two transition protocols (1:1 randomization).
  - o <u>Follow-up phase</u> (Week 2 to week 3): Subjects will return to their preclinical trial CSII regimen.

Figure 1: Study Design

192

193

194

195

196

197

198

199

200

201

202



## 3.4. Rationale for study design

205

206

207

208

209

210

211

212

213

214

215

216

217

218

219

220

221

222

223

224

225

and pharmacodynamics. Indeed, insulin degludec steady state concentration reaches 60% and 85% respectively at day 1 and 2, and 100% steady state is reached on day 3 from the first day of insulin degludec injection [12-13]. Therefore, 50% and 75% dose reduction proposed in the overlap transition strategy of the first 2 days will cover for the slow rise of insulin degludec concentration the first 2 days, and the 100% insulin pump discontinuation on day 3 will correspond to the time needed for insulin degludec to reach the steady state. This would reduce time spent in hyperglycemia post-CSII discontinuation. Rationale for blinded CGM: Since the primary outcome is time spent in hyperglycemia (CGM glucose >180 mg/dl), it is necessary to have CGM during randomized phase. Real-time CGM would interfere with the primary and secondary outcomes as patients will have ability to see CGM glucose trend and adjust insulin accordingly. Therefore, blinded CGM would be appropriate for this research protocol. In addition, the time in range (and percentage of hypoglycemia) also depends on person' ability to manage diabetes and therefore, baseline CGM will provide the data about time-in-range and time spent in hyper-and hypo-glycemia. The information from blinded CGM during run-in-phase will be useful for analysis of primary and secondary outcomes that will be adjusted for baseline CGM glucose metrics. Blood glucose fluctuations are greatest during the first week of insulin pump to MDI transition and therefore, 1 week CGM period is enough for comparison of primary and secondary outcomes between the groups.

The rationale behind the overlap protocol strategy is linked to insulin degludec pharmacokinetic

## 4. CLINICAL RESEARCH SITES

The study will be conducted at a single site, Barbara Davis Center for Diabetes.

# 228 **5. STUDY POPULATION:**

- We plan to enroll 34 participants with the expectation that 30 will be randomized and complete the
- study.
- 231 **5.1. Inclusion criteria**
- 232
- 233 1) Age  $\geq$ 18 years and  $\leq$  65 years
- 2) Patients with T1D diagnosed for at least 12 months
- 235 3) Point-of-care HbA1c levels between  $\geq 6.5\%$  and  $\leq 8.5\%$
- 236 4) Patients on CSII (any insulin pump) for at least past 6 months
- 5) Willing and able to wear a blinded CGM during the time of study period
- Willing to perform self-monitoring of blood glucose (SMBG) at least 4 times a day
- 239 7) Ability to provide informed consent before any trial-related activities
- Not willing to or plan any travel out of Colorado during the 3 weeks of study period
- 241 9) Willing to use insulin degludec in the morning once a day
- 242 **5.2.** Exclusion criteria
- 243
- 244 1) Age <18 years and > 65 years
- 245 2) HbA1c >8.5 % at screening
- 246 3) Less than 12 months of insulin treatment
- 247 4) Patients on 670G or Tandem Control IQ (Medtronic and Tandem Hybrid Closed-loop
- systems) and not willing use manual mode during the study period
- 249 5) Patients with T1D using any glucose lowering medications other than insulin
- 250 6) Pregnancy, breast feeding, and positive pregnancy test during screening

| 251 | (1) Women of childbearing age wanting to become pregnant or not using adequate |
|---|---|
| 252 | contraceptive measures |
| 253 | 8) Current or recent (< 2 weeks prior to visit 1) use of any steroidal medication, or anticipated |
| 254 | steroidal treatment, during the study period |
| 255 | 9) eGFR below 45 ml/min/1.73 m^2 using MDRD formula |
| 256 | 10) History of severe hypoglycemia in the previous 3 months |
| 257 | 11) History of diabetic ketoacidosis (DKA) requiring hospitalization in the past 3 months |
| 258 | 12) History of allergy to any form of insulin or its excipients |
| 259 | 13) History of allergy to adhesives |
| 260 | 14) Unwilling to use blinded CGM during the study period |
| 261 | 15) Unwilling to perform SMPG at least 4 times a day |
| 262 | 16) Known history of alcohol abuse or illicit drug use within 6 months prior to screening |
| 263 | 17) Use of investigational drugs within 5 half-lives prior to screening |
| 264 | 18) Participation to other study trials during the study period |
| 265 | 19) Elevated liver enzymes (AST and ALT) 3 times the upper limit of normal |
| 266 | 20) Hypoglycemia unawareness defined as GOLD score ≥4 [20] |
| 267 | 21) Any comorbidities or medical conditions that make a person unfit for the study at the |
| 268 | discretion of the investigators |
| 269 | 22) Anticipated travel across different time zones (difference greater than 4 hours) or |
| 270 | anticipated change in physical activities or diet at the discretion of the investigators. |
| 271 | |
| 272 | |

## 5.3. Withdrawal criteria

273

274

275

276

277

278

279

280

281

282

283

284

285

286

287

288

289

290

291

- Participation in this research is voluntary. Subjects may withdraw at will at any time. When withdrawing from the study, the participant should let the research team know that he/she wishes to withdraw. A participant may provide the research team with the reason(s) for leaving the study, but is not required to provide their reason.
- Participants will be withdrawn from the study if they become pregnant, actively try to
  become pregnant, develop an allergic reaction to insulin/adhesives, severe episodes of
  hypoglycemia/hyperglycemia, or at the judgement of investigators due to safety concerns,
  such as abnormality in laboratory exam results.
- After withdrawal, the participant will be given instructions on how to safely stop using study medications and, eventually, on how to correctly and safely return to the previous insulin regimen. Instructions are also given on who to contact if there are any questions or concerns that arise after study withdrawal.
- At the time of withdrawal, the research participant should let the research team know if
   he/she will allow the use of his/her health information and collected data by the researchers.

## 5.4. Subject replacement

- Subject replacement will occur only if withdrawal occurs before the one-week randomization phase. Subjects will not be replaced during the one-week randomized phase.
- 5.5. Rationale for study population
- In anticipation of screening failure or withdrawal or anticipated issues due to covid-19 pandemic, we plan to screen up to 40 subjects to have 30 complete the clinical trial.

294

#### 6. VISIT PROCEDURES:

## 6.1. Visit 1, week 0, day0, screening and blinded CGM insertion

- Subjects will attend a screening visit (Visit 1, week 0) in order to assess eligibility for the study.
- Before screening takes place, subjects will be provided with written information about the trial and the procedures involved. Subjects will be fully informed, both orally and in writing, about their responsibilities and rights while participating in the trial, as well as about possible advantages and disadvantages when participating in this trial. Subjects will have the opportunity to ask questions and have ample time to consider participation. The informed consent process will take place before the screening visit. Before signing the informed consent, the investigator will make sure that has full knowledge of the study processes, and the possibility to withdrawal at any time during the study.
- Subjects who wish to participate in the trial must sign and date the informed consent form for the trial before any trial-related procedures. All subjects will be provided with a copy of signed informed consent form.
- At screening, the subjects will be assigned a unique subject number, which will remain the same throughout the trial. The subject number will consist of 6 digits (the first 4 digits indicating the protocol number and the last 2 digits are unique for the subject).
- All subjects will undergo review of inclusion and exclusion criteria. If any inclusion criteria is answered 'no' or any exclusion criteria is answered 'yes', the subject is a screen failure, and no further assessment will take place.

- Patients will be told the importance of compliance in pre-set study visit time schedules.

  This will be true for both visits done at the BDC and phone call visits. After screening visit (visit 1, day 0), they will be asked to come at the BDC at visit 2 (day 7±1) and visit 3 (day 14±1). Furthermore, they must be compliant with phone call 1 (Week 1+24 hours; visit 2+24 hours), phone call 2 (Week 2+48 hours; P1+24 hours) and phone call 3 (day 21±1)
  - Point of care HbA1c and spot urine pregnancy test (for women in reproductive age group) will be done at the time of screening. A non-fasting blood will be drawn for complete metabolic panel (CMP).
  - If any clinical pathological condition is detected at physical examination, the investigator can decide, at his/her discretion, to withdraw the patient from the study.
  - For laboratory results such as CMP, "results pending" will be selected at Visit 1, week 0.
  - Please refer to Table 1 for a description of items to be performed at the screening visit.
    - All subjects will undergo GOLD questionnaire to exclude patients with hypoglycemia unawareness. Subjects with hypoglycemic unawareness defined as a GOLD score of ≥ 4
       [18] will be excluded.
    - All subjects will be assessed for ability to perform SMBG. Participants will be required to perform at least 4 SMBG daily using their own glucose meter; with at least one being in a fasted state, one pre-prandial and one 2-3 hours post-meal glucose value. In addition, participants will be required to check their blood glucose level if they have symptoms of hyperglycemia or hypoglycemia. We expect hyperglycemia during first 48-72 hours after randomization in group1 (standard of care transition). Therefore, SMBG requirements are

- necessary to select appropriate patients for this clinical trial for safety reasons. However,

  SMBG data will not be analyzed for primary or secondary endpoints.
  - All subjects will go through a quick review on diabetes self-management, including:
    - o Recognition of carbohydrates in commonly eaten foods
    - o Ability to count the carbohydrate content in typical portions of simple foods
    - o Ability to interpret a nutrition label for carbohydrate content
      - Preventing and treating hypoglycemia using carbohydrate-containing food and/or glucagon
  - All subjects will be instructed <u>NOT</u> to make any changes in the basal and bolus pump settings during run-in phase unless necessary for safety reasons (i.e. episodes of severe hypoglycemia or hyperglycemia) at discretion of investigators. If any therapy change will be necessary, it must be recorded.
  - Dexcom G6 will be inserted either on abdomen or upper arm depending on patient's preference and blinded at screening to analyze baseline CGM glucose metrics. The participants will not be able to see glucose values from the blinded CGM. All the subjects will be trained on function modalities of the blinded CGM. Dexcom G6 does not require calibration.
  - Patients on Medtronic 670 G (Medtronic hybrid closed-loop system where insulin pump delivers automatic basal rate based on Medtronic Guardian CGM glucose) will be instructed to use only pump (the Auto/ hybrid closed-loop mode will be disabled) because automatic insulin delivery can alter the primary objective of the study.

341

342

343

344

345

346

347

348

349

350

351

352

353

354

355

356

357

| 359 | • Patients using real time (rt) personal CGM (e.g. Freestyle Libre, Dexcom G4, Dexcom G5, |
|---|---|
| 360 | Medtronic Guardian Connect) will be screened for the study; however, they are not |
| 361 | allowed to use rt-CGM during the 2 weeks of the study (run-in-phase and randomization). |
| 362 | They can use rt-CGM during third week of the study while transitioning back to their own |
| 363 | insulin pump. |
| 364 | |
| 365 | 6.2. Screening Failure |
| 366 | Screening failure form must be completed. Resampling/ rescreening is not allowed if person failed |
| 367 | any of inclusion or exclusion criteria except for the laboratory criteria, where one-time rescreening |
| 368 | will be permitted at discretion of the investigator. |
| 369 | |
| 370 | 6.3. Visit 2, Week 1, Day 7±1, Randomization visit |
| 371 | <ul> <li>Blood glucose meter download and review of SMBG.</li> </ul> |
| 372 | <ul> <li>Subject's blinded CGM will be removed and downloaded.</li> </ul> |
| 373 | <ul> <li>Review of previous CMP lab data with patient.</li> </ul> |
| 374 | <ul> <li>Look for any local skin reaction at the site of previous CGM.</li> </ul> |
| 375 | • If glucose meter or CGM download shows a glucose value <54mg/dl, patient will be asked |
| 376 | if they experienced symptoms of hypoglycemia, if any assistance was required, and if there |
| 377 | were circumstances that possibly contributed to or resulted in hypoglycemia. |
| 378 | <ul> <li>Reporting of AE/ SAE if any</li> </ul> |
| 379 | <ul> <li>Exclusion criteria (after review of CMP laboratory and glucose meter data):</li> </ul> |

 $\circ$  AST/ALT > 3 times the upper limit of normal

| 381 | o eGFR <45 ml/min/1.73 m^2 using MDRD formula |
|---|---|
| 382 | o Abnormal laboratory results or allergic reaction at CGM site, which at the view of |
| 383 | investigator makes subject unsafe to continue the study. In that case, the |
| 384 | investigator has to explain the reason of his choice to the patient. |
| 385 | o Non-compliance defined as SMBG less than 4 times a day for at least 4 out of 7 |
| 386 | days and use of CGM less than 5 out of 7 days during the run-in-phase |
| 387 | <ul> <li>If no exclusion criteria was met, and the patient is still willing to continue the study,</li> </ul> |
| 388 | randomization process can start. |
| 389 | <ul> <li>Second, blinded CGM (Dexcom G6) will be inserted.</li> </ul> |
| 390 | ■ Subjects will receive 1 pen of insulin degludec U-100 and 1-2 pen of insulin aspart U-100 |
| 391 | depending on calculated insulin requirement during randomization phase. |
| 392 | <ul> <li>Diabetes self-management training including treatment of hypoglycemia and</li> </ul> |
| 393 | hyperglycemia will be reassessed. |
| 394 | <ul> <li>Subjects will be trained on the use of insulin pen and administration of correct dose of</li> </ul> |
| 395 | insulin degludec U-100 in the morning once a day and correct dose of insulin aspart U-100 |
| 396 | based on carbohydrate ratio and correction factor. |
| 397 | ■ Randomization |
| 398 | Subjects will be randomized equally into one of the two possible treatment arms. |
| 399 | o Group 1 (standard of care): subjects will stop using CSII on the randomization day, |
| 400 | and will start insulin degludec injection (1:1 dose conversion) once a day in the |
| 401 | morning. |

o Group 2 (overlap transition): Subjects will receive insulin degludec in full dose (1:1 dose conversion) at randomization, and CSII basal rate will be reduced by 50% during the first 24 hours of the transition and by 75% during 24 to 48 hours of the transition. CSII will be discontinued on day 3 of the transition.

The insulin degludec initiation and CSII basal reduction over 72 hours has been summarized in Table 2;

 Table 2: CSII changes and MDI initiation by randomization groups

| Randomization | Treatment<br>Change | V2 (Day 7±1) | P1 (V2+24 hours) | P2 (P1+24 hours) |
|---|---|---|---|---|
| Group 1(n=15) Standard of care | CSII | Discontinuation | | |
| | Insulin degludec | Once a day in the mor | rning (1:1 dose conversion) | |
| | Insulin aspart | Based on carbohydrat | e ratio and correction factor | ſ |
| Group 2(n=15) Overlap transition | | | 75% basal rate reduction | Discontinuation |
| | Insulin degludec | Once a day in the mor | rning (1:1 dose conversion) | |
| | Insulin aspart | No insulin aspart injections as patients will be using boluses through insulin pump | No insulin aspart<br>injections as patients<br>will be using boluses<br>through insulin pump | Insulin aspart injections based on carbohydrate ratio and correction factor |

- o Insulin degludec dose conversion guidance:
- On the day of randomization, CSII will be downloaded and information on average basal insulin for the last 3 days, carbohydrate ratio and correction factor will be recorded.
- The average basal insulin for last 3 days will be used to calculate insulin degludec U-100 starting dose. For example; average basal insulin during last 3 days of CSII is 20 units/day, the insulin degludec U-100 starting dose will be 20 units/day. The dose will be rounded up or down as needed. E.g. if patient's total daily dose is 32.4 units, it will be rounded to 32 units

- per day. All subjects will be instructed to use insulin degludec once a day in morning only.

  The first date of insulin deals declared will be given in the clinica at Wigit 2.
- The first dose of insulin degludec will be given in the clinics at Visit 2.

421

422

423

424

425

426

427

433

434

- The dose of insulin aspart will be based on patient's own carbohydrate ratio and correction factor. Carbohydrate ratio is defined as the number of carbohydrates covered by each unit of rapid acting insulin. Correction factor (aka insulin sensitivity factor) is defined as how much one unit of rapid acting insulin will drop blood glucose. For example; a patient with carbohydrate ratio of 1:15 and correction factor of 1:50 >150 will take 3 units if preprandial blood glucose is ~200 mg/dl for 30 grams of meal (2 units for 30 grams of carbs + 1 unit for correction). Subjects randomized to group 2 will be instructed to start insulin aspart 48 hours after randomization; i.e. when they disconnect their insulin pump.
- It is likely that patients randomized to standard-of-care group may experience

  hyperglycemia during first 48-72 hours. Therefore, both groups will be given a diary

  (Appendix 1) to record any correction made during the randomization phase to count extra

  insulin injections needed to correct blood glucose during first 72 hours.

## 432 6.4. Phone call 1 [P1, week 2, visit 2+24hrs] and phone call 2 [P2, week 2, P1+24hrs]

- As a safety measures, there will be 2 phone calls 24 and 48 hours after randomization, respectively.
- Phone call 1 (P1) will be done 24 hours (±6 hours in case if patient does not respond to first phone call) after visit 2.
- Phone call 2 (P2) will be done 24 hours (±6 hours in case if patient does not respond to first phone call) after P1.
- All subjects will be asked/assessed for

440 Any episodes of severe hyperglycemia requiring hospitalization or hypoglycemia 0 441 requiring third person' assistance. These events will be recorded as SAE and insulin 442 dose modification will be done at discretion of the investigator for safety reasons. 443 Correct insulin dose and administration will be reassessed. 444 Maintenance of glucose and insulin injection dairy. Any skin reaction at CGM site. 445 0 446 For Group 2 (overlap transition): 447 Instructions to change in basal rate (75% basal reduction) will be done at P1 Instructions for CSII discontinuation and initiation of insulin aspart based on 448 449 carbohydrate ratio and correction factor at P2 450 6.5. Visit 3, week 2, day 14±1: end of treatment 451 Blood glucose meter download and review of SMBG. 452 Subject's blinded CGM will be removed and downloaded. 453 Look for any local skin reaction at the site of CGM insertion. 454 Subjects will return all the remained study-related products (CGM device components, 455 insulin degludec and aspat pens, and any auxiliary supplies) 456 Report any AE/SAE if any. 457 Subjects will be transitioned back to their preclinical trial insulin pump regimen. The same 458 basal and bolus settings will be used as of preclinical trial insulin pump settings. However, 459 there may be changes made to basal and bolus insulin doses depending on blood glucose 460 control during the study period at the discretion of investigators. To reduce the risk of

| 461 | hypoglycemia, subjects will be advised to set a 50% temporary basal insulin rate for 24 hrs |
|---|---|
| 462 | following insulin degludec transition. |
| 463 | 6.6. Phone call 3, week 3, day 21±1: follow-up phone call and end of the study |
| 464 | • The intention of phone call 3 is to make sure that subjects are not experiencing major |
| 465 | hypoglycemia or hyperglycemia events. The study coordinator will make a phone call to |
| 466 | assist subjects if they require insulin dose adjustments. AE/ SAE will be recorded, if any, |
| 467 | during third week of clinical trial. However, they would not be a part of statistical analysis. |
| 468 | |
| 469 | |
| 470 | |
| 471 | |
| 472 | |
| 473 | |
| 474 | |
| 475 | |
| 476 | |
| 477 | |
| 478 | |
| 479 | |
| 480 | |
| 481 | |
| 482 | |

## 483 **6.7. Table 4: study visit outline**

| Period | Screening<br>and Run-<br>In-Phase | | Randomiza | tion | End of treatment | Follow-up |
|---|---|---|---|---|---|---|
| Visits | V1 | V2 | P1 | P2 | V3 | Р3 |
| Day/time from last visit | 0 | 7 | V2 + 24hrs | P1 +24hrs | 14 | 21 |
| Time window | | ±1 day | ±6hrs | ±6 hrs | ±1 day | ±1 day |
| Subject related info/assessment | | | | | | |
| Informed consent | X | | | | | |
| Inclusion/exclusion criteria | X | | | | | |
| Screen fail/withdrawal criteria | X | X | | | | |
| Demography and medical history | X | | | | | |
| Diabetes history | X | | | | | |
| GOLD questionnaire | X | | | | | |
| IDSS, and WPAI questionnaire | X | X | | | X | |
| Concomitant illnesses | X | | | | | |
| Review of current medications | X | | | | | |
| Vital signs | X | | | | | |
| BMI | X | | | | | |
| Physical examination | X | | | | | |
| Report AE/SAE | X | X | X | X | X | X |
| Trial material/steps | | | | | | |
| Dispensation of study drugs | X | X | | | | |
| SMBG and DSM education | X | | | | | |
| Glucose and insulin diary | | X | X | X | | |
| Blinded CGM insertion/training | X | X | | | | |
| Blinded CGM removal/download | | X | | | X | |
| SMBG profile | X | X | | | | |
| MDI initiation and training | | X | | | | |
| Randomization | | X | | | | |
| Transition back to CSII | | | | | X | |
| Compliance check | | X | | | | |
| Blood Draw | X | | | | X | |
| POC A1c, urine pregnancy test* | X | | | | | |
| CMP (blood sampling) | X | | | | | |

V1, V2, V3 stand respectively for visit 1, 2 3; P1, P2, P3 stand respectively for phone call 1, 2, 3

484

485

SMBG; self-monitoring of blood glucose, BMI; body mass index, DSM; diabetes self-

<sup>486</sup> management education, POC; point-of-care.

<sup>\*</sup>pregnancy test only for women in reproductive age.

490 491 6.8. Assessments for Safety: 492 The following safety assessments will be performed; 493 Time spent in CGM measured hypoglycemia (< 70 mg/dl) and time spent in hyperglycemia 494  $(\geq 250 \text{ mg/dl})$ 495 AE/SAE 496 Documented hypoglycemic episodes 497 Height, weight, vitals and physical examination 498 Baseline laboratory assessment 499 Hypoglycemia unawareness assessment (using GOLD questionnaire) 500 Pregnancy test at screening 501 6.9. Assessments for Efficacy: 502 The assessment for efficacy is time spent in CGM glucose time-in-range (min/ 24 hours, 70-180 503 mg/dl) during the 7 days of randomization period. 504 7. EVALUABILITY OF SUBJECTS: 505 The data for a subject with minimum of 5 out of 7 days of blinded CGM prior to randomization 506 and 5 out of 7 days of blinded CGM after randomization will be evaluable and included for the 507 analysis of primary and secondary objectives. 508 8. STATISTICAL CONSIDERATIONS: 509 8.1. Sample size calculation 510 In a study by Garg and colleagues, the subjects with T1D on MDI and blinded CGM for first 4 511

weeks of the study spent average of 8.8 hours/day (~528 min/ 24 hours) in CGM defined glucose

using CGM experienced average of 601 minutes (~10 hours/ day, IQR; 467-793 min) per 24 hours

above 180 mg/dl [21]. Similarly, in the recently published DIAMOND study, subjects on MDI

512

| of time spent in hyperglycemia [22]. We assume that subjects in standard of care group would |
|---|
| have more hyperglycemia than subjects in overlap transition group. Therefore, the expected CGM |
| hyperglycemia is $\sim 650$ minutes/24 hours in standard of care and $\sim 500$ minutes/24 hours in |
| overlap transition group with the differences in CGM glucose by150 minutes/day between the |
| groups. |
| This study is powered based on the primary endpoint, which is time spent in CGM-measured |
| glucose levels >180mg/dl (hyperglycemia). We have based the sample size on minimal relevant |
| differences between the two treatment groups, using a Type I error rate of 5% and a Type II error |
| rate of 20%. We hypothesize that the primary endpoint, time in minutes spent with glucose levels |
| >180 mg/dl, will be higher in the standard treatment group than in the experimental group (overlap |
| transition group), but we will use a two-sided test to assess differences in hyperglycemia by |
| treatment group. We hypothesize a standard deviation (SD) for time spent in hyperglycemia of |
| 140 minutes (2.3 hours, or $\sim$ 10% of the day) based on data from our clinic and previous |
| publications. We will have 80% power to detect a difference of 148.4 minutes (just under 2.5 |
| hours) between groups, which is a clinically meaningful difference in time spent hyperglycemia, |
| with a sample size of 15 participants completing the study per group (total N=30). We have also |
| calculated the detectable difference for larger SD estimates, in case the SD in the study population |
| is larger than in our clinic in general, and for 90% power. The effect sizes detectable with a final |
| sample size of 15 patients per group at 80% and 90% power are 1.06 and 1.23, respectively, for all |
| endpoints. |

| SD | Detectable difference (minutes) | Effect size | Power |
|---------|---------------------------------|-------------|-------|
| 140 min | 148.4 min | 1.06 | 80% |
| 160 min | 169.6 min | | 80% |
| 180 min | 190.8 min | | 80% |
| 140 min | 171.7 min | 1.23 | 90% |
| 160 min | 196.2 min | | 90% |
| 180 min | 220.8 min | | 90% |

538

539

Detectable differences in secondary CGM endpoints, including time in range (70-180 mg/dl) and time spent hypoglycemic (<70 mg/dl) have also been considered in our power analysis.

| Parameter | SD | Detectable difference | Power |
|---|---|---|---|
| | | (minutes) | |
| Time in range (70-180 mg/dl) | 160 min | 169.6 min | 80% |
| Time in range (70-180 mg/dl) | 180 min | 190.8 min | 80% |
| Time in range (70-180 mg/dl) | 200 min | 212.0 min | 80% |
| Time spent hypoglycemic (<70 mg/dl) | 45 min | 47.7 min | 80% |
| Time spent hypoglycemic (<70 mg/dl) | 60 min | 63.6 min | 80% |
| Time spent hypoglycemic (<70 mg/dl) | 75 min | 79.5 min | 80% |

540

541

## 8.2. Statistical Methods

- The proposed study includes two groups, one undergoing standard treatment and the other using a novel protocol of overlapping doses when transitioning from pump to MDI. Primary and secondary endpoints were described earlier.
- Study participants will be randomized using block randomization, but no stratification will be used since this is a small, single center trial.
- Our primary outcome is time spent hyperglycemic (CGM glucose values >180 mg/dl), which we will compared between randomized treatment groups (standard of care vs. novel overlap protocol)

during the transition from pump to MDI. We hypothesize that the time spent hyperglycemic will be reduced in the experimental group, using the novel overlap protocol, when compared to the standard treatment group. This hypothesis will be tested using a student's t-test to compare univariate differences between the standard care group and the experimental group for each of the outcomes. Secondary endpoints include time in range (70-180 mg/dl), time spent hypoglycemic (<70 mg/dl), frequency of severe hypoglycemia, number of correction boluses, and patient reported outcomes as defined on the page 7 of the protocol. Secondary endpoints will be examined using student's t-test to compare these outcomes univariately between the standard care and experimental groups. In a sensitivity analysis, CGM metrics will be evaluated in the first 72 hours vs entire 1 week as we expect that differences in hyperglycemia and time-in-range will be more pronounced between the two groups in the first 72 hours. For both primary and secondary endpoints, linear regression analysis will be used to examine outcomes by treatment group while adjusting for potential residual confounders, such as age and sex, which may not be fully addressed by randomization. All testing will be two-sided. The analysis will be conducted as an intention-to-treat analysis.

## 9. DATA HANDLING AND RECORD KEEPING:

- All data generated during the study will be retained by the investigator. Safety events will be reported to Colorado Multiple Institutional Review Board (COMIRB) in a timely manner as described under "Adverse Events".
- Data management is the responsibility of the investigator. All paper and electronic data will be saved in a de-identifiable manner. The data will be stored on BDC computers which are secured by the University of Colorado servers. The data will be accessible only

549

550

551

552

553

554

555

556

557

558

559

560

561

562

563

564

565

566

567

568

569

- by the study team and if transfer of data needed, appropriate measures, including encryption of data files will be used to ensure security and subject confidentiality.
- The records will be stored securely and kept for minimum of 10 years per the Standards
  Operating Procedures (SOP) of the University of Colorado [23].
- 575 [http://www.ucdenver.edu/research/Research%20Administration%20Documents/COMIRB 576 -Policy-and-Procedures-Document.pdf]

## 577 **10. ETHICS:**

578

579

580

581

582

583

584

585

586

587

588

- The trial will be conducted in compliance with this protocol, ICH GCP, the University of Colorado COMIRB research policy and in accordance with the Declaration of Helsinki [23-25].
- The clinical trial protocol, consent form and appropriate study documents will be submitted to COMIRB for the approval before the start of any study related activity.
  - Once the protocol is approved by the COMIRB, the study team will contact potential subjects from the BDC Adult clinic.
    - Before any trial-related activity, the investigator will give the subject verbal and written
      information about the trial and the procedures involved in a form that the subject can read
      and understand.
  - The subjects will be fully informed of their rights and responsibilities while participating in the trial as well as possible disadvantages of being treated with the trial products.
- The investigator will ensure the subject ample time to come to a decision whether to participate in the trial.

592 A voluntary signed and personally dated informed consent will be obtained from the 593 subject before any trial-related activity. 594 • The process of informed consent process will occur in a clinical research room located on 595 level 1, Barbara Davis Center for Diabetes Adult Clinic. The subject will sign the informed 596 consent process in the presence of the investigator and witness. The confidentiality and 597 HIPAA will be handled per the University of Colorado research policy. 598 11. STUDY SCHEDULE: 599 Trial registration: 4 weeks 600 Trial will be registered at Clinicaltrials.gov as soon as the study is funded. 601 Colorado Multiple Institutional Review Board (COMIRB): 2-3 months 602 The protocol, consent form, and appropriate trial materials will be submitted to COMIRB for 603 approval. 604 Planned duration of recruitment period: 7 months 605 Study duration from screening to the end of the study per subject- 3 weeks 606 Data cleaning and Statistical analysis: 2 months 607 Data presentation and publications: 6-12 months 608 12. STUDY DRUGS AND MATERIALS: 609 12.1. Study medications(s) / device(s) 610 Insulin: 611 Insulin degludec 100 units/ ml prefilled-pen 612 Insulin Aspart 100 units/ml prefilled-pen

Insulin degludec and Aspart will be provided by NovoNordisk.

Blinded CGM:

613

| 515 | <ul> <li>Dexcom G6 that will be blinded for the display. We would like to use Dexcom G6 as it</li> </ul> |
|---|---|
| 516 | does not require calibration and is most accurate CGM [26] amongst all marketed CGM. |
| 517 | Freestyle Libre is relatively inexpensive compared to Dexcom G6; however, Libre takes 12 |
| 518 | hours to warm- up and provide CGM values. The first 12 hours of CSII to MDI transition |
| 519 | is crucial for primary outcomes. |
| 520 | ■ Instructions to use Dexcom G6 |
| 521 | Insulin pump and pump related supplies would be patients own. Similarly, patients will use their |
| 522 | own blood glucose meter for SMBG. |
| 523 | 12.2. Packaging and labelling of study medication(s) |
| 524 | All the subjects will be provided sufficient study products including insulin pens, and pen needles. |
| 525 | Direction of use of insulin pen will be provided as outlines in the protocol. |
| 526 | Documentation of the study drugs/devices will be documented for each subject in accordance with |
| 527 | drug and device standard operating procedure of the Barbara Davis Center for Diabetes and the |
| 528 | University of Colorado Denver. |
| 529 | 12.3. Storage and drug accountability of study medication(s) |
| 530 | The drug (Insulin degludec and Aspart) will be stored according to approved label. The |
| 531 | temperature log will be monitored at the site and any temperature fluctuation will be reported as |
| 532 | deviation. |
| 533 | Subjects will be provided educational material(s) on direction of use of insulin and the storage. |
| 534 | Subjects will be instructed to store insulin in outer carton to protect from the light and cap should |
| 535 | be kept on the pen when not in use. Each insulin pump should be used within 26 days from the day |

of opening.

637 CGM (sensor and transmitters) will be stored per manufacturer' recommendation. 638 12.4. Auxiliary supply 639 The following will be supplied to study participants for the duration of clinical trial; 640 Needles for insulin pen, lancets, instruction for the use of insulin pens, instruction of CGM use and calibration. 641 642 13. CONCOMITANT ILLNESS(ES) AND MEDICATION(S) 643 Concomitant illness is any illness that is present at the start of the trial (i.e. at the first visit). For 644 each concomitant illness, date of onset, date of resolution or continuing, at a minimum, should be 645 recorded. 646 Concomitant medication is any medication other than the trial product(s) that are consumed during 647 the trial, including the screening and run-in periods. The information collected for each 648 concomitant medication includes, at a minimum, dosage, start date, stop date or continuing, and 649 indication. 650 Details of all concomitant illnesses and medication will be recorded at trial entry (i.e. at the first 651 visit). Any changes in concomitant medication must be recorded at Visit 6 at the time of 652 randomization. If the change influences the subject's eligibility to continue in the trial, the 653 investigator may withdraw the subject from the clinical trial. 654 **14. ADVERSE EVENTS:** 655 An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in 656 humans, whether considered drug related or not. AE can be unfavorable symptoms, sign 657 (abnormality on physical exam or laboratory findings) or disease temporarily associated with the 658 use of products whether or not related to the products.

659 Few examples (but not limited) of AEs are clinically significant worsening of concomitant illness, 660 a new illness, clinically significant radiological or laboratory abnormalities suggesting a disease or 661 organ toxicity. 662 The following three definitions are used when assessing an AE: 663 Severity assessment 664 Mild - no or transient symptoms, no interference with the subject's daily activities. **Moderate** - marked symptoms, moderate interference with the subject's daily 665 666 activities. 667 **Severe** - considerable interference with the subject's daily activities; unacceptable. 668 Causality assessment 669 The following terms are used when assessing the relationship between an AE and the 670 relevant study product(s): 671 Probable - Good reason and sufficient documentation to assume a causal 672 relationship. 673 **Possible** - A causal relationship is conceivable and cannot be dismissed. 674 **Unlikely** - The event is most likely related to etiology other than the study product. Final outcome of an AE 675 676 677 Recovered/resolved - The subject has fully recovered, or by medical or surgical

treatment, the condition has returned to the level observed at the first trial-related

activity after the subject signed the informed consent.

678

680 **Recovering/resolving** - The condition is improving and the subject is expected to 681 recover from the event. This term is only applicable if the subject has completed the 682 trial or has died from another AE. 683 Recovered/resolved with sequelae - The subject has recovered from the condition, 684 but with lasting effect due to a disease, injury, treatment or procedure. If a sequela 685 meets an SAE criterion, the AE must be reported as an SAE. 686 Not recovered/not resolved - The condition of the subject has not improved and 687 the symptoms are unchanged, or the outcome is not known. 688 **Fatal** - This term is only applicable if the subject died from a condition related to 689 the reported AE. Outcomes of other reported AEs in a subject before he/she died 690 should be assessed as "recovered/resolved", "recovering/resolving", "recovered/resolved with sequelae" or "not recovered/not resolved". An AE with 691 692 fatal outcome must be reported as an SAE. 693 **Unknown** - This term is only applicable if the subject is lost to follow-up. 694 Serious adverse event 695 An adverse event or suspected adverse reaction is considered "serious" if, in the view of the 696 investigator, it results in any of the following outcomes: 697 Results in death, or, 698 Is life-threatening, or, 699 Requires inpatient hospitalization or prolongation of existing hospitalization, or, 700 Results in persistent or significant disability/incapacity, or,

Is a congenital anomaly/birth defect,

- Is a medically important event that may not result in death, be life threatening or require
  hospitalization may be considered an SAE when based on appropriate medical judgement
  -they may jeopardize the subject and may require medical or surgical intervention to
  prevent one of the outcomes listed in the definition of SAE
- Suspected transmission of an infectious agent should be considered as an SAE.
- 707 Non-serious AE
- Any AE that does not fulfill the definition of SAE.
- 709 Medical event of special interest (MESI)
- A MESI is an event which, in the evaluation of safety, has a special focus. A MESI is an AE (SAE
- or non-serious AE) which fulfils one or more of the below defined MESI criteria.
- 712 Medication errors concerning trial products:
- 713 Administration of wrong drug
- 714 Wrong route of administration, such as intramuscular instead of subcutaneous
- 715 Accidental administration of a lower or higher dose than intended, however the
- 716 administered dose must deviate from the intended dose to an extent where clinical
- consequences for the trial subject were likely to happen as judged by the investigator,
- although not necessarily did happen.
- Overdose and missed insulin injection resulting in severe hypoglycemia or hyperglycemia are
- 720 considered as AE or SAE depending on severity.
- 721 Suspected Unexpected Serious Adverse Reactions (SUSAR)
- An unexpected adverse reaction (UAR) is an adverse reaction that is not consistent with the
- product information in the summary of product characteristics (SPC, i.e.US prescribing

- 724 information). The current version or any updated if available during the clinical trial for US
- prescribing information for study drugs will be used as SPC. If UAR is severe enough to define as
- 726 SAE is called as SUSAR.
- 727 <u>Technical complaint</u>
- A technical complaint is any written, electronic, or oral communication that alleges product
- 729 (medicine or device) defects. The technical complaint may be associated with an AE, but does not
- 730 concern the AE itself.
- 731 Reportable Device Issues
- AE and Unexpected Adverse Device Events (UADE) arising from the use of blinded CGM
- 733 (Dexcom G6) will be reported irrespective of severity, except in following cicumstances:
- The following device issues are anticipated and will not be reported unless the criteria for AE
- 735 reporting described above are met
- Component disconnections
- CGM sensors lasting fewer than 7 days
- CGM tape adherence issues
- Battery lifespan deficiency due to inadequate charging or extensive wireless
- 740 communication
- Intermittent device component disconnections/communication failures not leading to
- system replacement
- Device issues clearly addressed in the user guide manual that do not require additional
- 744 troubleshooting
- Skin reactions from CGM sensor placement that don't meet criteria for AE reporting

| $\overline{}$ | 1 | |
|---------------|----|---|
| | 71 | n |

760

761

763

765

766

767

768

**Safety Monitoring Officer** 

| 748 | A safety-monitoring officer (Aaron Michels, MD) will independently monitor the study, including |
|---|---|
| 749 | adverse events and study drug or device issues with potential to impact participant safety. A |
| 750 | monthly meeting will be held between study team and the safety officer to review any adverse |
| 751 | events. Following each safety review, a summary recommendation from the safety monitoring |
| 752 | officer will be collected. |
| 753 | Reporting and follow-up of adverse events |
| 754<br>755 | All events meeting the definition of an AE must be collected and reported. This includes events |
| 756 | from the first trial-related activity after the subject has signed the informed consent until the end of |
| 757 | the post-treatment follow-up period. |
| 758 | During each contact, the trained professional research associate will ask the subject about AEs and |
| 759 | technical complaints, for example by asking: "Have you experienced any problems since the last |

The investigator is responsible for reporting all AE to COMIRB within five business days per the

within 24 hours of the investigator's first knowledge of the SAE.

contact?". All AEs will be recorded by the investigator on an AE form. SAE will be recorded

University of Colorado Denver policy

764 (http://www.ucdenver.edu/research/Research%20Administration%20Documents/Unanticipated-Problem-

Reporting-Policy.doc). All non-severe and severe AE will be followed by till the end of the study

and will be reported to the COMIRB.

If a subject becomes pregnant during the study, the subject will be dropped from the study and

followed until the pregnancy outcomes. Pregnancy will be reported as AE (or SAE if fulfills the

- riteria of SAE) and it will be reported to the study sponsor (NovoNordisk). Pregnancy
- complications will be recorded as adverse events and if the infant has a congenital abnormality or
- birth defect, it will be reported and notified to the COMIRB and the sponsor.
- All SAE and SUSAR will be reported to NovoNordisk within 15 days from the investigator
- becoming aware of such adverse events. The following information will be provided to the
- sponsor; study name, patient identification (e.g. initials, sex, age), event (preferably a diagnosis),
- drug name, reporter identification (e.g. Name, or initials), causality, and outcome.

## 776 14.1. Precautions/over-dosage

- Insulin over or under dose can cause severe hypoglycemia or hypoglycemia. All subjects will be
- explained on the insulin dose and instructed on insulin pen use as a precautionary measures. The
- education on recognition of hypoglycemia or hyperglycemia and its treatment will be provided at
- 780 screening and as needed during the study.

## 781 **14.2 Risks and Discomforts**

- 782 a) Blood Drawing Risks
- 783 The risks of drawing blood from a vein include temporary discomfort from the needle stick
- 784 (common), bruising (common), excessive bleeding (unlikely), lightheadedness (rare), infection
- 785 (rare), and fainting (rare).
- 786 b) Fingerstick Risks (for A1c and finger stick glucose monitoring)
- 787 It may hurt when the lancet goes into a participant's finger but not for long. In about 1 in 10 cases,
- a small amount of bleeding under the skin will produce a bruise. A small scar may persist for
- several weeks. The risk of an infection is less than 1 in 1,000 people.
- 790 c) Related to CGM

Wearing sensors can cause adverse skin reactions such as pain at the site sensor insertion. The adhesive pads may cause skin erythema for 1 to 2 days or more. An allergic reaction to 1 or more parts of CGM devices may occur which can be mild, moderate, or severe (rare). In rare cases, an infection at the sensor site may occur. In rare cases, the sensor or needle may break inside the body and would require a minor surgical procedure to remove it. We will also screen out individuals with a history of serious skin reactions to adhesives.

d) Risk of Hypoglycemia (Low Blood Sugar)

As with any person with diabetes who uses insulin, there is always a risk of having low blood sugar (hypoglycemia). Symptoms of low blood sugar can include sweating, jitteriness, and not feeling well. There is also the possibility of fainting or seizures (convulsions), brain damage, or death with a very low blood sugar. Since we will be closely monitoring participants during this study, a serious low blood sugar is less likely to occur in any study participant. Even if a low blood sugar does occur, it usually goes away quickly with treatment (carbohydrates) that raises the blood sugar. A severe low blood sugar may require that a participant get an injection of glucagon and/or have emergency services to help raise his/her blood glucose level.

e) Risk of Hyperglycemia (High Blood Sugar)

Hyperglycemia usually does not cause many obvious symptoms, but participants may become thirsty, fatigued, or have a higher level of sugar in their urine. In severe cases of hyperglycemia, diabetic ketoacidosis (DKA) or coma may occur. Hyperglycemia leading to DKA can lead to renal failure (kidney failure), cardiac arrhythmia (irregular heartbeat), myocardial infarction (heart attack), rhabdomyolysis (muscle breakdown), and even death. A serious effect from

812 hyperglycemia is not expected to occur in any study participant, as we will be monitoring blood 813 glucose levels frequently. 814 f) Psychosocial Questionnaires 815 Answering questionnaires about thoughts, concerns, and distress related to diabetes and general 816 quality of life assessments may result in undesired thought processes and/or emotions. These 817 feelings may be transitory, recurrent, or permanent though most risks are minimal/transitory. 818 g) Unknown Risks 819 In any study, there may be additional risks that we do not know about at this time. This is not 820 likely but is always a possibility. If we become aware of any new risks, participants will be told 821 about them. They will be able to decide if they want to continue to participate in this study. If a 822 treatment or procedure has increased risks because it was not done according to study procedures 823 due to error, participants will be informed, and the necessary steps will be taken to care for them. 824 h) Confidentiality 825 There is a risk of a breach in confidentiality. Thus, a confidential subject database will be 826 established to maintain study data. Data will be entered into REDCap (Research Electronic Data 827 Capture). REDCap is an internal secure, computerized database system at the University of 828 Colorado Denver. This system allows data entry, survey/questionnaire building, data exportation 829 to statistical packages, and is HIPAA compliant. Each subject will be assigned an identification 830 number, which will be used to code and identify all of that subject's records. This will avoid the 831 continual use of subject names. REDCap surveys can be sent to study participants via e-mail for 832 direct input into the database. All study data will be locked in the PIs' offices and all relevant 833 computer study files will be input on staff computers, which are password protected and contain

encryption software. Data storage will be on a secured server maintained by the University of Colorado. The server is backed up nightly and a copy of the back-up file is kept off site in a secure facility. Data access will be limited to study personnel. Study results may be presented in the form of posters, abstracts, oral presentations, or publications at academic meetings or in journals. In all forms of study result reporting, subject identification will not be disclosed. A study subject may access his/her protected health information at any time by requesting said information in writing of the investigator. The investigative team has been trained in IRB and HIPAA compliance issues and will maintain confidentiality and protect health information. The above-stated procedures have been highly effective in preventing breaches of patient confidentiality for the prior and current research studies in which the PI has been and continues to be involved.

## **15. PUBLICATION PLAN:**

We plan to present the data at ADA and/or EASD depending on the time of completion of the analysis. The study will be published in a peer-reviewed scientific journal. The data will be publically assessable through clinicaltrial.gov. Authorship of publications will be in accordance with the Uniform Requirements of the International Committee of Medical Journal Editors.

## **16. REFERENCES**

- Atkinson MA, Eisenbarth GS, Michels AW. Type 1 diabetes. Lancet. 2014;383:69 82.PMID: 23890997
- Shah VN, Moser EG, Blau A, Dhingra M, Garg SK. The future of basal insulin. Diabetes
   Technol Ther. 2013 Sep;15(9):727-32.
- 3. Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs
  DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes
  treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes
  Care. 2015 Jun;38(6):971-8
- Maahs D, Horton LA, Chase HP. The use of insulin pumps in outh with Type 1 diabetes.
   Diabetes Technol Ther. 2010 Jun; 12(Suppl 1): S-59–S-65.
- Wong JC, Boyle C, DiMeglio LA, et al. Evaluation of Pump Discontinuation and
   Associated Factors in the T1D Exchange Clinic Registry. *Journal of Diabetes Science* and Technology. 2017;11(2):224-232. doi:10.1177/1932296816663963.
- 6. **Shah, V.N**., et al., Human factors associated with insulin pump and continuous glucose monitor discontinuation among adults with type 1 diabetes. Diabetes Technol Ther, 2016. 18(S1): p. A18.
- 7. Allison Blass. Taking a Pump Vacation, diabetes mine, 2017. Available at <a href="https://www.healthline.com/diabetesmine/taking-a-pump-vacation">https://www.healthline.com/diabetesmine/taking-a-pump-vacation</a>
- 875 8. Kurtzhals P, Heise T, Strauss HM, et al. Multi-hexamer formation is the underlying basis 876 for the ultra-long glucose-lowering effect of insulin degludec. Diabetologia. 877 2011;54(suppl 1):S426.
- 9. Jonassen I, Havelund S, Hoeg-Jensen T, et al. Design of the novel protraction mechanism of insulin degludec, an ultra-long-acting basal insulin. Pharm Res. 2012;29:2104–2114. doi: 10.1007/s11095-012-0739-z.
- 10. Heise T, Heinemann L. Rapid and long-acting analogues as an approach to improve insulin therapy: an evidence-based medicine assessment..Curr Pharm Des. 2001 Sep; 7(14):1303-25.

- 11. Lane W, Bailey TS, Gerety G, et al. Effect of Insulin Degludec vs Insulin Glargine U100 on Hypoglycemia in Patients with Type 1 Diabetes: The SWITCH 1 Randomized Clinical Trial. *JAMA*. 2017; 318(1):33-44. doi:10.1001/jama.2017.7115.
  - 12. Coester H-V, Heise T, Nosek L, et al. Steady state is reached within 2 to 3 days of once-daily administration of ultra-long-acting insulin degludec. Diabetologia. 2012;55 (suppl 1):373.
- 13. Haahr H, Heise T. A review of the pharmacological properties of insulin degludec and their clinical relevance. Clin Pharmacokinet 2014;53:787-800
  - 14. Kaufman FR. Insulin Pumps and Continuous glucose monitoring- A user's guide to effective diabetes management. Editor 1. Publisher American Diabetes Association.
- 894 15. Walsh J, Roberts R. Pumping insulin. Third edition. Torrey Pine Press.
- 895 16. Bolderman KM. Putting your patients on the pump. American diabetes Association.
- 17. Chase P. Understanding Insulin pumps and continuous glucose monitors. 1<sup>st</sup> edition.
   Children's Diabetes Foundation, Denver, CO.
  - 18. Polonsky WH, Fisher L, Hessler D, Edelman SV. Development of a New Measure for Assessing Insulin Delivery Device Satisfaction in Patients with Type 1 and Type 2 Diabetes. Diabetes Technol Ther 2015;17:773-9.
  - 19. Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics 1993;4:353-65.
    - 20. Gold AE, MacLeod KM, Frier BM: Frequency of severe hypoglycemia in patients with type 1 diabetes and impaired awareness of hypoglycemia. Diabetes Care 17:697–703, 1994
  - 21. Garg SK, Voelmle MK, Beatson CR, Miller HA, Crew LB, Freson BJ, Hazenfield RM. Use of continuous glucose monitoring in subjects with type 1 diabetes on multiple daily injections versus continuous subcutaneous insulin infusion therapy: a prospective 6-month study. Diabetes Care. 2011 Mar;34(3):574-9.
- 22. Beck RW, Riddlesworth TD, Ruedy KJ et al for DIAMOND Study Group. Effect of
   initiating use of an insulin pump in adults with type 1 diabetes using multiple daily

888

889

892

893

898

899

900

901

902

903

904

905

906

907

908

| 912 | insulin injections and continuous glucose monitoring (DIAMOND): a multicentre, |
|---|---|
| 913 | randomised controlled trial. Lancet Diabetes Endocrinol. 2017 Sep;5(9):700-708. |
| 914 | 23. University of Colorado Denver. Colorado Multiple Institutional Review Board |
| 915 | (COMIRB) policies and procedures. Available at |
| 916 | http://www.ucdenver.edu/research/research%20administration%20documents/comirb- |
| 917 | policy-and-procedures-document.pdf. Accessed on March 19, 2018 |
| 918 | 24. World Medical Association. World Medical Association Declaration of Helsinki: ethical |
| 919 | principles for medical research involving human subjects. JAMA. 2013;310(20):2191- |
| 920 | 2194. |
| 921 | 25. International Conference on Harmonisation. ICH Harmonized Tripartite Guideline. Good |
| 922 | clinical Practice 01 May 1996. |
| 923 | https://www.ich.org/fileadmin/Public_Web_Site/ICH_Products/Guidelines/Efficacy/E6/ |
| 924 | E6_R1_Guideline.pdf. Accessed on March 19, 2018 |
| 925 | 26. Shah VN, Laffel LM, Wadwa RP, Garg SK. Performance of a Factory-Calibrated Real- |
| 926 | Time Continuous Glucose Monitoring System Utilizing an Automated Sensor |
| 927 | Applicator. Diabetes Technol Ther. 2018 Jun;20(6):428-433. |
| 928 | |
| 929 | |
| 930 | |
| 931 | |
| 932 | |
| 933 | |
| 934 | |
| 935 | |
| 936 | |
| 937 | |
| 938 | |
| 939 | |
| 940 | |

**Appendix 1:** Glucose and Insulin Dose Diary

Glucose and Insulin dose Logbook

Study protocol noStudy personnel name and contactPhone- email

| Time 12am 1 2 3 4 5 6 7 8 9 10 11 12p 1 2 3 4 5 BG Readings | 6 7 | 8 | 9 | 10 | 11 |
|---|---|---|---|---|---|
| Carbs (Grams) Carb boluses Correction bolus Total Insulin Aspart dose Additional Details: Breakfast Lunch Dinner | | | | | <u>+</u><br>+ |
| Carb boluses Correction bolus Total Insulin Aspart dose Additional Details: Breakfast Lunch Dinner | | | | | + |
| Correction bolus Cotal Insulin Aspart dose Additional Details: Breakfast Lunch Dinner | | | | | |
| bolus Total Insulin Aspart dose Additional Details: Breakfast Lunch Dinner | | | | | - 1 |
| otal Insulin spart dose Additional Details: Breakfast Lunch Dinner | | | | | |
| Additional Details: Breakfast Lunch Dinner | | | | | |
| Time Food Description amount Carb griss Time Food Description amount Carb griss Time Food Des | pariation | omour | nf | Cork | gms |
| | scription | amour | nt | Carr | gms |
| | | | + | | |
| | | | + | | |
| Morning Snacks Afternoon Snacks Evening Snacks | | | <u> </u> | | |
| | | | t | | |

# 952 Table: Summary of protocol changes and rationale.

| Revisions | Rationale |
|---|---|
| Email address change (page 1) | Due to domain change at CU Anschutz, email |
| Eman address change (page 1) | address of the protocol PI was changed |
| Exclusion criteria 4. (page 10) | Tandem Control IQ is a HCL system that is approved by the US FDA for T1D in December 2019. Therefore, it is added in the exclusion criteria. |
| Section 5.5 (page 12). Total number of patients required for screening are increased from 34 to 40. | Due to covid related institutional closure and restrictions, we lost data for 1 patient, 1 patient withdrew from study and 4 screen failed, we increased screening sample size to have 30 patients complete the entire study to have adequate power. |
| Insulin degludec dose conversion guidance (page 18). | A line is added to have clarification that if total insulin dose in last 3 day is rounded for calculation of insulin degludec. E.g. is patient's total daily dose is 32.4, it is rounded to 32.0 and if 32.7, it is rounded to 33.0 units per day. |
| Sample size calculation (Page 24 and 25) | Typographical errors were corrected on page 24 and 25. |
| Statistical Methods (Page 26) | Sensitivity analysis of CGM metrics in the first 72 hours vs entire 1 week is added. This is because we expect the differences in hyperglycemia to be more pronounced in the first 72 hours. |
| Secondary endpoint 4: there was a typographic mistake (page 7) | As stated on page 19, we intended to collect correction boluses information during first 72 hours only. |